CLINICAL TRIAL: NCT04469179
Title: A Phase 1B, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study of SAB-185 in Ambulatory Subjects With COVID-19
Brief Title: Safety, Tolerability, and Pharmacokinetics of SAB-185 in Ambulatory Participants With COVID-19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SAb Biotherapeutics, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency); Joint Program Executive Office (JPEO) Chemical, Biological, Radiological, and Nuclear Defense (CBRND) Enabling Biotechnologies (EB) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAB-185-102
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: COVID-19; SARS-CoV2
MeSH Terms: conditions — COVID-19 | interventions — SAB-185; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): 10mg/kg SAB-185 in normal (0.9%) saline; concentration 4mg/mL (0.4%)
  Interventions: Biological: SAB-185
- Cohort 2 (Experimental): 25mg/kg SAB-185 in normal (0.9%) saline; concentration 20mg/mL (2%)
  Interventions: Biological: SAB-185
- Cohort 3 (Experimental): 50mg/kg SAB-185 in normal (0.9%) saline; concentration 20mg/mL (2%)
  Interventions: Biological: SAB-185
- Placebo (Placebo Comparator): Normal (0.9%) saline in approximately the same volume as each cohort in the experimental drug arm.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: SAB-185 — SAB-185 is a purified human immunoglobulin G (hIgG) designed to specifically bind to Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) viruses. SAB-185 is purified from the plasma of immunized Tc bovines that were immunized initially (vaccinations 1 and 2) with a plasmid DNA (pDNA) vaccine that expresses wild-type SARS-CoV-2 spike protein, followed by additional immunizations (vaccinations 3 and beyond) with a recombinant spike protein from SARS-CoV-2 produced in insect cells. The purified hIgG is a sterile liquid formulated in 10 mM glutamic acid monosodium salt, 262 mM D-sorbitol, 0.05 mg/mL Tween 80, pH 5.5. The drug product will be administered intravenously and will be diluted in saline per the clinical protocol.
  Other Names: Anti-SARS-CoV-2 Human Immunoglobulin Intravenous (Tc bovine-derived)
  Arms: Cohort 1; Cohort 2; Cohort 3
Other: Normal Saline — Normal (0.9%) saline in approximately the same volume as each cohort in the experimental drug arm.
  Arms: Placebo

SUMMARY:
: Coronavirus disease 2019 (COVID-19) is an infectious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). SAB Biotherapeutics has developed SAB-185, an Anti-SARS-CoV-2 Human Immunoglobulin Intravenous (transchromosomic [Tc] bovine-derived), as a potential therapeutic to treat COVID-19. This study will evaluate the safety, immunogenicity, and pharmacokinetics of SAB-185 in ambulatory participants with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria for inclusion:

1. 18-60 years of age
2. Positive for presence of SARS-CoV-2 on NP or OP swab by FDA-authorized RT-PCR test within seven days prior to infusion
3. At least one current symptom of COVID-19, onset within seven days prior to infusion:

   * Fever or chills
   * Cough
   * Shortness of breath or difficulty breathing
   * Fatigue
   * Muscle or body aches
   * Headache
   * New loss of taste or smell
   * Sore throat
   * Congestion or runny nose
   * Nausea or vomiting
   * Diarrhea
4. Able to understand the study and comply with all study procedures
5. Agrees not to participate in any other trial of an investigational product during the study period
6. Willing and able to provide written informed consent prior to the start of any study related activities
7. If female, meets at least one of the following reproductive risk criteria

   * Post-menopausal for at least 12 months
   * Use of one or more of the following highly effective contraceptive methods for at least 90 days following the last dose of study product: combined estrogen and progestogen containing or progestogen-only hormonal contraception, intrauterine device (IUD), intrauterine hormone-releasing system, surgical bilateral tubal occlusion
   * Vasectomized sole sexual partner who has received medical assessment of the surgical success
8. Male and female subjects agree to sexual abstinence (refraining from heterosexual intercourse for at least 90 days following the last dose of study product) if not using birth control or condoms for males.

Exclusion Criteria:

Subjects who meet any of the criteria of severe or higher COVID-19 will be excluded from the study:

* Dyspnea at rest
* Respiratory rate > 30 breaths per minute
* SpO2 ≤ 93% on room air
* Heart rate ≥ 125 beats per minute
* Respiratory distress or respiratory failure.
* Evidence of critical illness

  1. Female subjects with positive pregnancy test, breastfeeding, or planning to become pregnant/breastfeed during the study period.
  2. Hospitalization or need for hospitalization for any cause
  3. Treatment or participation in another clinical trial of any other investigational agent within 30 days prior to enrollment.
  4. Use of other drugs that, in the opinion of the investigator, could complicate analysis of SAB-185.
  5. Subjects with the following risk factors:
* Compromised immune system including confirmed diagnosis of current cancer under treatment, inherited deficiencies of the immune system, immune suppressing medication, or other conditions causing leukopenia or neutropenia
* Known autoimmune condition requiring therapy more intensive than intermittent non-steroidal anti-inflammatories in the prior 6 months (for example: rheumatoid arthritis, lupus, inflammatory bowel disease)
* Chronic respiratory disease including COPD, emphysema, cystic fibrosis, pulmonary hypertension, or other chronic condition that requires the routine use of supplemental oxygen
* Chronic asthma requiring the use of oral steroids or hospitalization in the last six months
* Renal failure or renal insufficiency requiring dialysis
* Congestive heart failure or significant atherosclerotic disease (coronary artery disease or peripheral vascular disease) 6. Receipt of pooled immunoglobulin or plasma in past 30 days 7. Any other underlying medical (cardiac, liver, renal, neurological, respiratory) or psychiatric condition that in the view of the investigator would preclude use of SAB-185 8. Known IgA deficiency or previous allergic reaction to intravenous immunoglobin (IVIG)/subcutaneous immunoglobin (SCIG) 9. Positive for hepatitis B virus surface antigen, hepatitis C virus antibody, or HIV antibody by medical history 10. History of allergy, anaphylaxis, or severe reaction to beef products (including milk and gelatin).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Having Adverse Events | 29 Days
  Incidence and severity of other adverse events and severe adverse events (SAE)
Number of Participants Having Transfusion-Related Adverse Events | 29 Days
  transfusion-related adverse events

SECONDARY OUTCOMES:
Number of Participants Having Adverse Events | 90 Days
  Incidence and severity of adverse events and SAEs from Screening through Study Day 90
Assesment of the PD of SAB-185 administered intravenously | 90 Days
  Measurement of SARS CoV-2 neutralizing (PRNT80) antibody titers from screening through Study Day 90
Immune response elicited by SAB-185 | 90 Days
  Measurement of Rheumatoid factor through day 90
Concentration of subject anti-SAB-185 antibodies elicited by SAB-185 | 90 Days
  Measurement of anti-SAB-185 antibodies through screening day 90
Incidence of SARS-CoV-2 in oropharyngeal (OP) or nasopharyngeal (NP) swab specimens | 29 Days
  Incidence of SARS-CoV-2 in swab specimens as measured by quantitative RT-PCR through Study Day 29
Level of SARS-CoV-2 in oropharyngeal (OP) or nasopharyngeal (NP) swab specimens | 29 Days
  Level of SARS-CoV-2 in swab specimens as measured by quantitative RT-PCR through Study Day 29

CONTACTS AND LOCATIONS:
Overall Officials: David Hoover, MD, Principal Investigator — ICON GPHS
Locations (3):
- United States (3):
  - Quantum Clinical Trials, Miami Beach, Florida
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Sanford Health, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the published article, after deidentification (test, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication and ending 36 months following article publication
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343